CLINICAL TRIAL: NCT02614833
Title: AIPAC (Active Immunotherapy PAClitaxel): A Multicentre, Phase IIb, Randomised,Double Blind, Placebo-controlled Study in Hormone Receptor-positive Metastatic Breast Carcinoma Patients Receiving IMP321 (LAG-3Ig Fusion Protein) or Placebo as Adjunctive to a Standard Chemotherapy Treatment Regimen of Paclitaxel
Brief Title: IMP321 (Eftilagimod Alpha) as Adjunctive to a Standard Chemotherapy Paclitaxel Metastatic Breast Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Immutep S.A.S. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMP321 P011
Record Dates: First submitted 2015-11-05; First posted 2015-11-25 (Estimated); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Adenocarcinoma Breast Stage IV
Keywords: Hormone receptor positive
MeSH Terms: interventions — soluble LAG-3 protein, human; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel + IMP321 at the RPTD (Experimental): The chemo-immunotherapy phase consists of 6 cycles of 4 weeks. Patient will receive weekly paclitaxel at Days 1, 8 and 15 with adjunctive treatment of study agent, either IMP321, on Days 2 and 16 of each 4-week cycle. After completion of the 6-cycle chemo-immunotherapy phase, responding or stable patients will receive study agent (IMP321) every 4 weeks during the maintenance phase for an additional period of up to 12 injections
  Interventions: Biological: IMP321 (eftilagimod alpha); Drug: Paclitaxel
- Comparator: Paclitaxel + Placebo (Active Comparator): The chemo-immunotherapy phase consists of 6 cycles of 4 weeks. Patient will receive weekly paclitaxel at Days 1, 8 and 15 with adjunctive treatment of study agent, placebo, on Days 2 and 16 of each 4-week cycle. After completion of the 6-cycle chemo-immunotherapy phase, responding or stable patients will receive study agent (placebo) every 4 weeks during the maintenance phase for an additional period of up to 12 injections
  Interventions: Drug: Placebo; Drug: Paclitaxel

INTERVENTIONS:
Biological: IMP321 (eftilagimod alpha) — In the placebo-controlled, double-blind randomisation stage, paclitaxel + IMP321 at the RPTD will be compared to paclitaxel + placebo
  Arms: Paclitaxel + IMP321 at the RPTD
Drug: Placebo — In the placebo-controlled, double-blind randomisation stage, paclitaxel + placebo will be compared to paclitaxel + IMP321 at the RPTD
  Arms: Comparator: Paclitaxel + Placebo
Drug: Paclitaxel — Paclitaxel will be given in both treatment arms (classified as Non IMP)

SUMMARY:
The proposed Phase IIb clinical study aims to investigate the safety and efficacy of the active immunotherapy IMP321 in combination (adjunctive) with paclitaxel chemotherapy in patients with hormone receptor-positive metastatic breast cancer.

DETAILED DESCRIPTION:
This is a multicentre, placebo-controlled, double-blind, 1:1 randomised Phase IIb study in female hormone receptor-positive metastatic breast cancer patients. The study comprises of two stages.

Stage 1 is the open-label, safety run-in stage consisting of cohort 1 and 2 to confirm the (RPTD) of IMP321 in combination with paclitaxel.

Stage 2 is placebo-controlled, double-blind randomisation stage, paclitaxel + IMP321 at the RPTD will be compared to paclitaxel + placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give written informed consent and to comply with the protocol
2. Metastatic oestrogen receptor positive and/or progesterone receptor positive breast adenocarcinoma, histologically proven by biopsy of the primary tumour and/or metastasis
3. Female of age 18 years or above
4. Patients who are indicated to received first line chemotherapy with weekly paclitaxel
5. Evidence of measurable disease as defined by Response Evaluation Criteria version 1.1

6 Laboratory criteria: haematology and biochemistry results within the limits normally expected for the patient population.

Exclusion Criteria:

1. Prior chemotherapy for metastatic breast adenocarcinoma
2. Disease-free interval of less than twelve months from the last dose of adjuvant chemotherapy
3. Inflammatory carcinoma
4. Candidate for treatment with trastuzumab (or other Her2/neu targeted agents)
5. Systemic chemotherapy, radiation therapy or any other investigational agent within 4 weeks, endocrine therapy within 1 week prior to first dose of study treatment or CDK4/6 inhibitors within 5 times half-life (acc.to SPC) prior to first dose of study treatment and until completion of study treatment
6. Symptomatic known cerebral and/or leptomeningeal metastases
7. Serious intercurrent infection
8. Evidence of severe or uncontrolled cardiac disease (NYHA III-IV) within 6 months prior to first dose of study treatment
9. Active acute or chronic infection
10. Active autoimmune disease requiring immunosuppressive therapy
11. Previous malignancies within the last three years other than breast carcinoma
12. Patients with prior organ or stem cell transplantation
13. Any condition requiring continuous systemic treatment with either corticosteroids or other immunosuppressive medications within 4 weeks prior to first dose of study treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2015-12; Primary Completion 2020-03 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Stage 1 to determine the recommended phase two dose for the randomised phase | Up to 12 months
Assessment of Progression-Free Survival (PFS) | Up to 37 month

SECONDARY OUTCOMES:
Assessment of the safety and tolerability of IMP321 as compared to placebo | Up to 19 months
Assessment of the overall survival (OS) | Up to 48 month
Stage 1: Evaluation of the pharmacokinetic e.g. Peak Plasma Concentration [Cmax] | Up to 12 months
Assessment of the change in quality of life (QOL) | Up to 37 months
Evaluation of the time to next treatment | Up to 37 months
Evaluation of objective response rate (ORR) | Up to 37 months
Evaluation of stable disease | Up to 37 months

OTHER OUTCOMES:
Stage 1: assessment of Immuno-monitoring in a defined subset of 60 patients during the randomised stage | Up to 37 months

CONTACTS AND LOCATIONS:
Overall Officials: Immutep S.A.S, Study Director — Immutep S.A.S.
Locations (29):
- Belgium (8):
  - AZ Sint-Jan Burgge-Oostende, Bruges
  - Cliniques universitaires Saint-Luc - Institut Roi Albert II - Cancérologie et Hématologie Oncologie clinique, Brussels
  - AZ Sint-Maarten, Duffel
  - Universitair Ziekenhuis Antwerpen Breast and Gynecological Oncology Unit, Edegem
  - UZ Leuven, campus Gasthuisberg Department of General Medical Oncology and Multidisciplinary Breast Centre, Leuven
  - Clinique Sainte-Elisabeth, Namur
  - AZ Nikolass, Sint-Niklaas
  - GZA Ziekenhuizen campus Sint-Augustinus Oncologische Research, Wilrijk
- France (3):
  - Institut Curie / Centre René Huguenin, Saint-Cloud
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - Institut Claudius Regaud - IUC Toulouse - Oncopôle, Toulouse
- Germany (5):
  - KEM- Brustzentrum der Kliniken Essen-Mitte, Essen
  - Onkologische Gemeinschaftspraxis am Bethanien-Krankenhaus Centrum für Hämatologie und Onkologie, Frankfurt
  - NCT - Nationales Centrum für Tumorerkrankungen, Heidelberg
  - UFKT - Universitäts-Frauenklinik Tübingen, Tübingen
  - UFU - Universitätsfrauenklinik Ulm, Ulm
- Hungary (2):
  - Szent Margit Kórház Onkológiai Osztály, Budapest
  - MH Egészségügyi Központ Onkológiai Osztály, Budapest
- Netherlands (7):
  - VU University Medical Center, Amsterdam
  - Zuyderland MC, Geleen
  - UMCG Medisch Centrum Groningen, Groningen
  - HMC Antoniushove, Leidschendam
  - MUMC Medical Oncology department, Maastricht
  - Erasmus MC, Rotterdam
  - VieCuri Medisch Centrum, Venlo
- Kierownik Oddziału Onkologii i Radioterapii Szpital Morski im. PCK w Gdyni, Gdynia, Poland
- United Kingdom (3):
  - St James' Institute of Oncology, Leeds, West Yorkshire
  - The Christie NHS Foundation Trust The Christie Clinic - Medical Oncology, Manchester
  - Nottingham University Hospitals NHS Trust, Nottingham